CLINICAL TRIAL: NCT00792194
Title: Improvement of Aerobic Capacity in Cystic Fibrosis Patients With a One-year Home Training Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007-A01452-51
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Exercise training; Home training; Aerobic capacity
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- training group (Experimental): supervised training program 3 times a week with coach.
  Interventions: Other: Exercise training
- group without training (No Intervention): a control group, where subjects are asked to continue their normal daily activities and physiotherapy regime.

INTERVENTIONS:
Other: Exercise training — Subjects will be randomised in two groups:
  a control group, where subjects are asked to continue their normal daily activities and physiotherapy regime.
  a training group, where subjects are asked to exercise three times a week, whenever they want during the day.
  Other Names: no applicable
  Arms: training group

SUMMARY:
Life expectancy of patients with cystic fibrosis has improved dramatically the last few years. Respiratory complications remain the main contributory factor to the morbidity and mortality associated with the disease. Exercise tolerance is reduced as the disease progresses, and peak aerobic capacity seems to be linked with survival. Regular physical activity has positive benefits, including a better body image, an improvement of pulmonary function, of exercise capacity and a possible improvement of quality of life.But because of the considerable variability of the subjects, exercise programs should be tailored to individual needs, and easy included in their cumbersome treatment routines and professional activities. In the cystic fibrosis center of Strasbourg we are able to propose to the patients a one-year physical exercise program, partly supervised with coaches, at home. Electronically braked cycle ergometer and heart rate monitoring system are at patients disposal, for one year, at home. Thus, patients can choose, during the day, the best moment to work out .Subjects will be randomised in two groups:1. a control group, where subjects are asked to continue their normal daily activities and physiotherapy regime.2. a training group, where subjects are asked to exercise three times a week. For the training group, three times a week, patients will train for 30 minutes. Heart rate will be continuously monitored and send to the medical staff every week-end . A correction of exercise intensity, if needed, is weekly proposed to maintain a maximal training efficiency, and coaches can help them, if necessary. For the two groups, quality of life will be measured with a disease-specific questionnaire (CFQ14+) (Henry, 1998, Quittner, 2000), and a generic questionnaire (SF 36) (Gee, 2002) before the program, and after 6 and 12 months. After a one year training program, and compared to the control group, we should expected an improvement in aerobic capacity and peak oxygen consumption, both associated with improved prognosis in cystic fibrosis. We also expected to observe an improvement in quality of life measurement, shorter hospital stays and fewer exacerbations. With this kind of program, we also would like to improve the degree of adherence in daily life exercise.

DETAILED DESCRIPTION:
We hope that regular contact with the coaches or the medical staff will provide self-confidence. Thus, patients will probably be more able to choose a physical activity which will be enjoyable, shared with others (family, friends), and give real benefits in term of health status.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman with cystic fibrosis whose diagnosis was documented on clinical history and a test for detecting genetic or sweat test positive
* Patient who signed the informed consent (or parents for patients minors)
* Elderly aged 15 and over
* Patient affiliated with a social security
* Patient against non-cardiac indication of physical
* Patient in stable condition on a respirator with a higher FEV to 1000 ml
* In the case of insulin-dependent diabetes, it must be balanced
* Patient had been informed of the results of the medical examination
* Women of childbearing age have achieved a pregnancy test on urine negative.

Exclusion Criteria:

* Diabetic patient unbalanced known cardiac pathology
* Patient on transplant list
* Patient major protected
* Patient under guardianship or trusteeship
* Safeguard patient justice

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changing the criteria for assessing aerobic capacity: Variations in VO2 max. | 4 years

SECONDARY OUTCOMES:
Assess the impact of retraining at home Going on the frequency of exacerbations, length of hospital stays, daily energy expenditure. Assess the impact of retraining at home | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: LONSDORFER Evelyne, MD, Principal Investigator — not affiliated
Locations (1):
- CHRU, Hôpital Civile, Service de Physiologie et Explorations Fonctionnelles, Strasbourg, France